CLINICAL TRIAL: NCT06316791
Title: Exploratory Clinical Study of CNCT19 Anti CD19 Cell Therapy in the Treatment of Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001007
Record Dates: First submitted 2024-03-04; First posted 2024-03-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: CNCT19; CD19-directed CAR-T cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered before the investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Autologous 2nd generation CD19-directed CAR-T cells, infusion intravenously.

SUMMARY:
Exploratory clinical study of CNCT19 anti CD19 cell therapy in the treatment of refractory autoimmune diseases,To evaluate the safety and tolerability of CNCT19 in patients with refractory systemic lupus erythematosus (lupus nephritis, immune thrombocytopenia), refractory ANCA-associated vasculitis, and refractory dermatomyositis on the basis of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The enrolled subjects or their legal representatives signed informed consent form;
2. age range: 18-70 years (including 18 and 70 years), male or female;
3. Subjects with refractory systemic lupus erythematosus (lupus nephritis, immune thrombocytopenia) : Diagnosed with systemic lupus erythematosus according to American College of Rheumatology (ACR) criteria, accompanied by lupus nephritis (SLE-LN) or immune thrombocytopenia (SLE-ITP) and receiving standard treatment;

   1. Subjects with Refractory Systemic Lupus Erythematosus (Lupus Nephritis): Active and biopsy-confirmed proliferative lupus nephritis grade III or IV or simple grade V alone according to 2003 ISN/RPS criteria. Active renal disease was defined as a urine protein: creatinine ratio > 1.0 or proteinuria > 3.5 grams/day.
   2. Subjects with refractory systemic lupus erythematosus (thrombocytopenia): At least two consecutive blood routine examinations showed that platelet was lower than 50x109/L; Blood cell morphology of peripheral blood smear was normal. The spleen is generally not enlarged; The morphological characteristics of bone marrow cells were megakaryocytic increase or normal, accompanied by maturation disorder. Platelet count > 10 x10^9 / L.
4. Subjects with refractory ANCA-associated vasculitis: diagnosis of ANCA glomerulonephritis (GN) or vasculitis based on the 2013 American Chapel Hill Consensus Conference definition of AAV ;

   * Relapsed or refractory AAV requiring treatment with cyclophosphamide or rituximab
   * Newly diagnosed or recurrent AAV--, defined as accumulation of at least one major organ (e.g., kidney, lung, heart) requiring induction therapy with cyclophosphamide or rituximab;
   * Anti-PR3 or anti-MPO positive (current or history);
5. Subjects with Refractory Dermatomyositis: Refractory MDA5-positive dermatomyositis is defined as active disease and meets the following conditions: adequate corticosteroid therapy (greater than two to four weeks of conventional corticosteroid therapy or intolerance to such therapy) and/or

   * Use of ≥ 1 conventional immunosuppressive agent (eg, methotrexate, azathioprine, tacrolimus, cyclosporine, mycophenolate mofetil, IVIG, anti-TNF, or rituximab) at a reasonable dose and duration (greater than two to four weeks or intolerance to therapy);
   * Treatment with IVIG or cyclophosphamide for two to four weeks.
6. Women of childbearing potential must have a negative blood pregnancy test 7 days prior to trial conditioning therapy; any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for at least 1 year following reinfusion of CNCT19 CAR-T cells. Childbearing potential, in the judgment of the investigator, is biologically capable of bearing a living baby and sexually active. Female patients who were not of childbearing potential (ie, met at least 1 of the following criteria):

   * Hysterectomy or oophorectomy, or
   * Medically confirmed ovarian failure, or medically confirmed postmenopausal (cessation of menses for at least 12 consecutive months in the absence of pathological or physiological causes).
7. Adequate organ function according to the following criteria:

   * Aspartate aminotransferase (AST) ≤ 3 times of upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) ≤ 3 times ULN;
   * Total serum bilirubin ≤ 2 times ULN unless the patient has documented Gilbert's syndrome; patients with Gilbert's syndrome who have bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included;
   * Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula), Patients with lupus nephritis may relax the conditions appropriately according to the judgment of the investigator;
   * Must have minimal pulmonary reserve and oxygen saturation > 91% in a nonoxygenated state;
   * Lymphocyte count > 0.4 × 109/L.

Exclusion Criteria:

1. Patients with severe active central nervous system (CNS) lupus, including seizures, psychosis, cerebrovascular accident or CNS vasculitis requiring therapeutic intervention within 60 days after baseline;
2. Dialysis patients;
3. Pregnancy or lactation;
4. Concomitant uncontrollable infection (e.g., sepsis, bacteremia, fungemia, uncontrolled pulmonary infection, etc.);
5. Hepatitis B surface antigen (HBsAg) positive and hepatitis C (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive, syphilis (TP) positive;
6. Major surgery that was assessed as unsuitable by the investigator within 4 weeks before screening;
7. Patient's heart meets any of the following:

   * Left ventricular ejection fraction (LVEF) ≤ 45%;
   * New York Heart Association (NYHA) Class III or IV congestive heart failure or active cardiac disease;
   * Serious arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia);
   * QTc interval ≥ 450 ms for males and ≥ 470 ms for females (QTcB = QT/RR1/2);
   * Myocardial infarction, bypass surgery or stent surgery within 6 months prior to the study;
   * Other cardiac diseases that are not suitable for the study as judged by the investigator;
8. Received live vaccine within 6 weeks prior to screening.
9. Participation in other interventional clinical studies within 3 months prior to cell infusion, treatment with an active experimental drug, or intentional participation in another clinical trial or treatment outside of that specified by the protocol throughout the study period.
10. Patients with a history of epilepsy or other active central nervous system diseases;
11. Known hypersensitivity to the ingredients of the preparation used in the test;
12. Prior treatment with CAR-T cells.
13. Other conditions that the investigator considers inappropriate for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects Experiencing Treatment-Emergent Adverse Events（TEAE） | Up to 1 year after CNCT19 infusion
  Evaluate the type, frequency, severity of adverse events, and abnormal laboratory test values; Evaluate the frequency and severity of adverse events related to CNCT19.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1 year after CNCT19 infusion
  The time from the CNCT19 Cell Injection infusion to death due to any cause
SELENA-SLEDAI | Up to 1 year after CNCT19 infusion
  0 to 4 is basically no disease activity;5 to 9 is light activity;10 to 14 is moderate activity;≥15 is considered heavy activity.
The proportion of subjects who achieved glucocorticoids/immunosuppressant free and subjects who achieved low-dose glucocorticoids application during the main study period | Up to 1 year after CNCT19 infusion
To evaluate disease related biomarkers | Up to 1 year after CNCT19 infusion
  Levels of anti nuclear antibodies, anti double stranded DNA antibodies, anti small ribosomal nucleoprotein antibodies
To evaluate disease related biomarkers | Up to 1 year after CNCT19 infusion
  Levels of anti C1q antibodies
To evaluate disease related biomarkers | Up to 1 year after CNCT19 infusion
  Levels of anti cardiolipin antibodies (IgG, IgM, IgA)
To evaluate disease related biomarkers | Up to 1 year after CNCT19 infusion
  Levels of anti MDA5 antibody (melanoma differentiation associated gene 5) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Shengyun Liu, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China